CLINICAL TRIAL: NCT04399772
Title: A COgNitive FuncTional Therapy+ Pathway Versus an Interdisciplinary Pain Management Pathway for Patients With Severe Chronic Low Back Pain (CONFeTTI Trial): a Randomized Controlled Trial of a Combined Physical/Psychological Intervention
Brief Title: COgNitive FuncTional Therapy+ for Chronic Low Back paIn
Acronym: CONFeTTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Curtin University (Other); Manchester Metropolitan University (Other)
Responsible Party: Principal Investigator, Henrik Bjarke Vægter, Professor in Physiotherapy, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 69712
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Chronic Low-back Pain
Keywords: Low back pain; Cognitive Functional Therapy; Interdisciplinary pain management; RCT; Disability
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: This study is a patient-blinded 2-arm randomized controlled trial with a parallel group design and 1:1 group allocation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study has ethical approval that the patients involved are not aware that there is a difference between the two treatment strategies in the study. Patient masking in this study is done to ensure that included patients are as representative as possible.
  The randomization sequence is distributed and stored in sealed opaque envelopes handled only by an independent study secretary who has no other involvement in the trial. All outcome measurements are completed via an electronic questionnaire system sent via personal links to the patients' official digital inbox, e-Boks (used by public hospitals, municipalities and other institutions to send official documents to citizens of Denmark). The researcher responsible for the statistical analyzes are blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Functional Therapy+ pathway (Experimental): Treatment is performed by a CFT trained physiotherapists and a psychologist in the Pain Center. Patients receive max 10 consultations over 3 months. The first two sessions is combined with the physiotherapist and psychologist who investigates potential maintaining factors for pain and disability in the patient's everyday life. Remaining sessions are run by the physiotherapist, and the treatment is individually tailored to the needs of the individual patient, aiming to provide the patient with skills in dealing with his / her own situation via information, reflection, change of movement and training of functions and physical level. The psychologist provide extra support for 2-3 sessions to reinforce the physiotherapist work.The ethical committee made blinding conditional on a possibility of usual care after CFT+ if: the patient does not feel ready to stop treatment AND analgesic treatment is inappropriate OR the social situation is problematic OR significant psychological distress.
  Interventions: Behavioral: Cognitive Functional Therapy+ pathway
- Interdisciplinary pain management pathway (Active Comparator): Treatment at the Interdisciplinary University Pain Center are based on elements from cognitive-behavioral therapy, Acceptance and Commitment Therapy, and Mindfulness-Based Stress Reduction programs.
  Treatment can be diverse, but based on an individual assessment it consists of a combination of (1) medical treatment with a specialist pain consultant+specialist pain nurse (ie, individual adjustment of analgesics to improve effect and reduce side effects) AND (2) one or more of the following: individual consultations with a specialist pain psychologist, physiotherapist or social worker with cognitive-behavioral therapy training as well as participation in a group program with relaxation therapy, acceptance and commitment therapy or standardized mindfulness-based stress reduction programs. On average patients in the pain center receives 9-10 sessions.
  Interventions: Behavioral: Interdisciplinary pain management pathway

INTERVENTIONS:
Behavioral: Cognitive Functional Therapy+ pathway — The CFT+ intervention comprises 4 main components: (1) making sense of pain: context-based patient education focusing on the multidimensional nature of pain and disability, while reducing the threat of structural damage and correcting unhelpful beliefs; (2) exposure with control: graded exposure to painful, feared, or avoided activities with body relaxation; (3) lifestyle changes: encouraged to perform physical activity based on preference and taught strategies to manage stress and poor sleep, (4) focus on coping strategies in life and how these strategies influence the current situation.
  After CFT+, patients can be offered the comparator pathway should that be clinically indicated from these criteria: the patient does not feel ready to stop treatment AND Analgesic treatment is inappropriate OR Social situation is problematic OR Significantly psychological distress that requires further treatment by psychologist. This decision is based on a multidisciplinary team conference.
  Arms: Cognitive Functional Therapy+ pathway
Behavioral: Interdisciplinary pain management pathway — Treatment at the Interdisciplinary University Pain Center are based on elements from cognitive-behavioral therapy, Acceptance and Commitment Therapy, and Mindfulness-Based Stress Reduction programs.
  Individualized combination of (1) medical treatment with a specialist pain consultant+specialist pain nurse (ie, individual adjustment of analgesics to improve effect and reduce side effects), (2) one or more of the following: individual consultations with a specialist pain psychologist, physiotherapist or social worker with cognitive-behavioral therapy training as well as participation in a group program with relaxation therapy, acceptance and commitment therapy or standardized mindfulness-based stress reduction programs.
  Arms: Interdisciplinary pain management pathway

SUMMARY:
This study is a patient-blinded 2-arm randomized controlled trial (RCT) assessing the effectiveness (in the short and long term) as well as total healthcare costs of a CFT+ (a combined physiotherapist/psychologist intervention) pathway compared with interdisciplinary pain management pathway (usual care) for patients with chronic low back pain referred to interdisciplinary pain treatment.

The primary aim of this pragmatic randomized controlled trial (RCT) is to investigate if a physiotherapy-led CFT pathway that includes psychologist support (CFT+) with the option of additional usual care (if needed) is superior to the currently recommended interdisciplinary pain management pathway (usual care) in reducing disability at 12 months in patients with severe cLBP. In addition, an economic evaluation will investigate total health care costs of the two pathways at 12 months.

In addition the study will explore changes in pain intensity, quality of life, thoughts and beliefs about back pain, and analgesic consumption in patients randomized to the CFT+ pathway compared with patients randomized to the interdisciplinary pain management pathway.

DETAILED DESCRIPTION:
Evidence suggests that chronic low back pain (LBP) is a multidimensional biopsychosocial problem including various contributing factors, such as negative pain cognitions, pain-related fear and emotional distress, avoidant and protective movement behaviors,and unhelpful lifestyle factors such as activity avoidance and sleep problems. Current guidelines recommend that patients with chronic LBP who do not benefit from primary care treatment should be referred to interdisciplinary pain rehabilitation in secondary care settings. However, such treatments are often expensive, not easily accessible, and have only modest effects.

Cognitive Functional Therapy (CFT) is a newer physiotherapeutic treatment approach for patients with chronic low back pain, involving all important elements for the individual patient. Physical factors are handled via change in pain-provoking movement patterns. Psychological factors are handled in relation to fear, avoidance behaviour, catastrophization, stress, anxiety, depression and negative thoughts. Lifestyle factors are addressed in relation to physical inactivity and sleep problems. The approach is individualized and provides the patient with opportunities for action in relation to his or her own situation via information, reflection, change of movement and training of functions and physical level.

CFT has been shown to reduce fear and worry in patients with chronic low back pain compared to other interventions, and the effect of CFT alone on patients with severe chronic low back pain has been recently investigated in an observational pilot study (without randomization) in our Pain Center (publication attached in link). In this study, we found a good and clinically relevant effect of CFT compared to standard treatment in a University Hospital Interdisciplinary Pain Center. In the pilot study, we noted that there were barriers to optimal treatment engagement for some patients (e.g. lack of motivation), and that several patients with high levels of psychological distress had limited benefits. Inclusion of early psychologist support to assist in promoting behavioral change and directly target deeper behavioral strategies could potentially improve patient adherence to the CFT intervention.

This fully-powered randomized controlled study compares effectiveness of this physiotherapeutic intervention including psychologist support (CFT+) pathway with effectiveness of interdisciplinary pain treatment (recommended care) pathway in patients with severe chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75 years referred to interdisciplinary pain management at the Pain Center
* Adequate Danish language skills
* • Chronic low back pain (pain in the area between the 12th rib and buttock crease lasting more than 6 months)
* Low back pain self-reported as significant contributor to daily disability (Yes/No)
* Low back pain intensity > 4 on 0-10 numerical rating scale
* Provide consent that data collected via questionnaires and registries can be used for research purposes

Exclusion Criteria:

* Previously attended an interdisciplinary pain management program
* Wheel chair bound
* Suicidal ideation - evaluated using Patient Health Questionnaire-9 (Item 9 has to be answered "never")
* Self-reported former/ present addictive drug or alcohol behavior
* Self-reported current pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2020-09-27 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Pain-related disability during the last 7 days | Change from baseline to 12 months
  Proportion of patients who have an improvement of 8 points or more on the Oswestry Disability Index (ODI) at 12 months. The ODI assesses pain-related disability within the last 7 days, asking patients to reflect on their ability to manage their everyday life despite their back pain for these domains: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and travelling. Each domain is scored on a 0-5 scale. The index is calculated by dividing the summed score by the total possible score multiplied by 100 and expressed as a percentage with 100 representing the greatest disability.

SECONDARY OUTCOMES:
Trajectory of Pain-related disability during the last 7 days | Assessed after 0, 3, 6, 9, and 12 months
  Assessed with the Oswestry Disability Index (ODI) that asks patients to choose statements that reflect their ability to manage their everyday life despite their back pain for these domains: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and travelling. Each domain is scored on a 0-5 scale. The index is calculated by dividing the summed score by the total possible score multiplied by 100 and expressed as a percentage with 100 representing the greatest disability.
Average pain intensity during the last 24 hours | Assessed at 0, 3, 6, 9, and 12 months
  Assessed by asking the participants about the level of average pain during the last 24 hours on a 11 point rating scale, ranging from 0-10 (0 = "no pain" and 10 = "worst pain") using the 5th item from the Brief Pain Inventory Short Form. A lower score indicates lower pain intensity.
Health-related quality of life | Assessed at 0, 3 and 12 months
  Measured by European Quality of Life 5 Dimensions (EQ-5D-3L) and the Visual Analogue Scale (EQ-VAS).
  For the 5 dimensions the EQ5D-3L asks the participants to rate their ability for each domain (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), respectively on a 1-3 Verbal Rating Scale, a score of 1 indicating no problems/severity, and a score of 3 indicating extreme problems/severity. The EQ-VAS asks the participant to rate their overall health 'today' on a 0-100 VAS. A higher score indicates a better quality of life.
Level of pain catastrophization | Assessed at 0, 3 and 12 months
  Measured by the Pain Catastrophizing Scale; asking participants to indicate the degree to which they experienced each of 13 thoughts or feelings when experiencing pain, on a 5-point Likert scale with 0 = not at all and 4 = all the time. The score is 0 to 52 with a higher score indicating a high level of pain catastrophizing.
Level of patient enablement | Assessed at 0, 3 and 12 months
  Measured by the Patient Enablement Instrument for Back Pain; asking participants to indicate on a 11 point rating scale, ranging from 0-10 (0 = "to a very low degree" and 10 = "to a very high degree") the degree to which they during the past week were able to 1) Cope with life, 2) Understand your back problem, 3) Cope with your back problem, 4) Keep your back healthy, 5) Feel confident about your health, and 6) Help yourself.
Economical evaluation | Assessed at 12 months
  The economic evaluation of the RCT will estimate the cost per quality adjusted life year (QALY) gained from the CFT+ intervention, compared to interdisciplinary pain program treatment. The economic analyses will utilize the EQ5D data collected during the trial for the utility weights, and total healthcare costs will be obtained from linking the trial data to Danish registries.
Analgesics | Assessed at 0, 3 and 12 months
  Use of analgesics (opioids, NSAIDs, Paracetamol, TCA) within the last week reported by the patient by a Yes or No answer.
Adverse reactions | Assessed at 3, 6, 9 and 12 months
  Assessed by asking the patient to report the occurence of any serious adverse reactions or adverse reactions during the last 3 months.
The Patient Global Impression of Change | Assessed at 3, 6, 9 and 12 months
  The Patient Global Impression of Change (PGIC) scale using Likert scale responses (1=much worse, 2=worse, 3=a little worse, 4=neither worse nor better, 5=a little better, 6=better, 7=much better).

OTHER OUTCOMES:
Depression (for patient description) | Baseline
  Depressive symptoms are assessed using the Patient Health Questionnaire-9 (PHQ-9). Nine items related to the core symptoms of depression are assessed on a 4-point Likert scale, ranging from 0 = 'not at all' to 3 = 'nearly every day', getting a score between 0 and 27 with a higher score indicating higher depression severity.
Anxiety (for patient description) | Baseline
  Anxiety symptoms are assessed with the Generalized Anxiety Disorder-7 (GAD-7) questionnaire. Seven items are assessed on a 4-point Likert scale, ranging from 0 = 'not at all' to 3 = 'nearly every day', getting a score between 0 and 21 with a higher score indicating higher anxiety severity.
Kinesiophobia (for patient description) | Baseline
  Kinesiophobia is assessed using the 17-item Tampa Scale of Kinesiophobia (TSK) questionnaire. Each of the 17 items is rated on a 4-point Likert scale with 1 = 'strongly disagree' and 4 = 'strongly agree', getting a score between 17 and 68 with a higher score indicating higher levels of fear of movement/kinesiophobia
Pain distribution (for patient description) | Baseline
  Self-reported drawing on body chart

CONTACTS AND LOCATIONS:
Overall Officials: Henrik B Vægter, PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Pain Center, University Hospital Odense, Odense, Funen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vaegter HB, Johansen JV, Sopina L, Smith A, Kent P, Fuglsang KS, Pedersen JF, Schutze R, O'Sullivan P, Handberg G, Fatoye F, Ussing K, Stegemejer I, Thorlund JB. A Cognitive Functional Therapy+ Pathway Versus an Interdisciplinary Pain Management Pathway for Patients With Severe Chronic Low Back Pain (CONFeTTI Trial): Protocol for a Pragmatic Randomized Controlled Trial. Phys Ther. 2021 Sep 1;101(9):pzab132. doi: 10.1093/ptj/pzab132. PMID 34003285
- See also: CFT pilot study in the Pain Center — https://journals.lww.com/painrpts/pages/articleviewer.aspx?year=2020&issue=02000&article=00004&type=Fulltext